CLINICAL TRIAL: NCT03881566
Title: Study of Usefulness of Presepsin as Early Detective Marker of Sepsis in Immunodeficiency ICU Patients
Brief Title: Presepsin as Detective Marker of Sepsis in Immunodeficiency ICU Patients
Acronym: PREICU
Status: Completed | Type: Observational
Sponsor: Jongmin Lee (Other)
Responsible Party: Sponsor-Investigator, Jongmin Lee, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: PRESEPSIN_IMMUNODIFFICIENCY
Record Dates: First submitted 2019-03-09; First posted 2019-03-19 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Sepsis; Immune Deficiency
MeSH Terms: conditions — Sepsis; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma, Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Immunocompetent sepsis patients: Sepsis patients without HIV infection (all stages), neutropenia (neutrophil count < 1 × 109/L), exposure to glucocorticoids (> 0.5 mg/kg for > 30 d) and/or immunosuppressive or cytotoxic medications, solid organ transplantation, allogeneic or autologous stem cell transplantation, hematological malignancy, or solid tumor.
- Immunocompromised sepsis patients: Sepsis patients with HIV infection (all stages), neutropenia (neutrophil count < 1 × 109/L), exposure to glucocorticoids (> 0.5 mg/kg for > 30 d) and/or immunosuppressive or cytotoxic medications, solid organ transplantation, allogeneic or autologous stem cell transplantation, hematological malignancy, or solid tumor.
- Patients without sepsis: Patients who admitted intensive care unit without sepsis

SUMMARY:
This is an observational study to evaluate the diagnostic and prognostic value of presepsin in the critically-ill immunocompromise patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 19 years
* Appropriate clinical data to enable classification into sepsis
* Written informed consent by the patient or legally authorized representative
* Critical illness consistent with sepsis, to be enrolled within 24 hours of presentation

Exclusion Criteria:

* No informed consent
* A patient who is judged to be unable to make a voluntary decision by understanding information about this research due to cognitive vulnerability

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with presentation to ICU with critical illness compatible with sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (ROC-AUC) of the Plasma Presepsin Concentration for Discriminating Between immunocompetent and immunocompromised patients. | up to 7 days
  For the analysis, plasma presepsin levels on Day 0 will be used. Sepsis was made on Day 7 or day of discharge. ROC-AUC of presepsin for discriminating between immunocompromised and immunocompetent patients is compared to that of procalcitonin.

SECONDARY OUTCOMES:
survival at ICU discharge or day 28 after enrollment | 28 days
  For the analysis, we will evaluate the association between presepsin and survival at ICU discharge or day 28 after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jongmin Lee, M.D., Study Director — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea